CLINICAL TRIAL: NCT05397197
Title: A Longitudinal Study of the Impact of Moderate Preterm Birth on Cortical and Subcortical Processing of Speech Sounds and Vocabulary Acquisition
Brief Title: Impact of Moderate Preterm Birth on Vocabulary Acquisition
Acronym: BABYLANG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-24; 2021-A02615-36 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2022-05-21; First posted 2022-05-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Premature Birth
Keywords: speech acquisition; prematurity; sounds processing; EEG
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Longitudinal follow-up (Other): Follow-up of children at 40 weeks of corrected age for all children and then regularly until 24 months
  Interventions: Other: Electroencephalography

INTERVENTIONS:
Other: Electroencephalography — experimental task, neuropsychological evaluation, clinical exam

SUMMARY:
Children born prematurely may present a neurodevelopmental disorder with a language delay diagnosed as early as 2-3 years of age. This situation is not uncommon: each year in France, approximately 35,000 children are born between 32 and 36 weeks of amenorrhea.

In our most recent work, we have shown that moderate premature infants show an attenuated cortical response to a vowel change, suggesting a deficit in the cortical encoding of vowels. This work needs to be continued in order to better understand syllable encoding and identify the neuroplasticity mechanisms underlying early speech encoding.

The identification of markers to predict language development is essential for the screening of these children at risk of language delay. These children could thus benefit from early adapted care even before the appearance of language deficits.

ELIGIBILITY:
Inclusion Criteria:

* Infants born prematurely (32-36 weeks gestational age, GA) or at term (40-2 weeks gestational age, GA)
* Birth weight appropriate to gestational age determined by WHO growth charts (weight, height, head circumference)
* Normal clinical examination at inclusion.
* Written informed consent obtained from both parents (or single parent if single parent)
* Infant with at least one parent who speaks and understands fluent French
* Infant is affiliated with the social security system
* Infant whose parents reside in Marseille

Exclusion Criteria:

* Neonatal distress (Apgar score < 7)
* Hypoxic and ischemic encephalopathy
* Perinatal acidosis
* Intrauterine growth retardation
* Brain injury (such as intraventricular or periventricular hemorrhage, periventricular leukomalacia)
* Cerebral congenital malformations
* Neonatal epilepsy
* Any condition that in the opinion of the investigator would not be compatible with the conduct of this study
* Abnormal hearing test performed as part of the child's routine care at birth,

Ages: 0 Days to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2028-10-19 (Estimated); Study Completion 2030-10-19 (Estimated)

PRIMARY OUTCOMES:
Study the impact of moderate prematurity on speech encoding characteristics development | 40 amenorrhea weeks
  Latency and amplitude of cortical and subcortical auditory evoked potentials in response to syllables, measured by Electroencephalography
Study the impact of moderate prematurity on speech encoding characteristics development | 3 months
  Latency and amplitude of cortical and subcortical auditory evoked potentials in response to syllables, measured by Electroencephalography
Study the impact of moderate prematurity on speech encoding characteristics development | 6 months
  Latency and amplitude of cortical and subcortical auditory evoked potentials in response to syllables, measured by Electroencephalography
Study the impact of moderate prematurity on speech encoding characteristics development | 10 months
  Latency and amplitude of cortical and subcortical auditory evoked potentials in response to syllables, measured by Electroencephalography
Study the impact of moderate prematurity on speech encoding characteristics development | 18 months
  Latency and amplitude of cortical and subcortical auditory evoked potentials in response to syllables , measured by Electroencephalography
Study the impact of moderate prematurity on speech encoding characteristics development | 24 months
  Latency and amplitude of cortical and subcortical auditory evoked potentials in response to syllables , measured by Electroencephalography

CONTACTS AND LOCATIONS:
Overall Officials: Francois Cremieux, Study Director — AP-HM
Locations (1):
- Service de Neuropédiatrie, Marseille, France

IPD SHARING:
Plan to Share IPD: No